CLINICAL TRIAL: NCT06067256
Title: A Multicentre, Prospective, Open-label, Non-comparative Study to Evaluate Menstrual Bleeding Typology, Tolerability, and Compliance During a Monophasic Hormonal Contraceptive Treatment With Norgestimate + Ethinylestradiol in Italy.
Brief Title: A Multicentre, Prospective, Open-label, Non-comparative Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: EFFI2021/01
Record Dates: First submitted 2023-09-28; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Contraception
Keywords: Female contraception
MeSH Terms: interventions — Contraceptive Agents, Female

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Female Contraceptive — Effimia® exerts its action by means of a gonadotropin suppression mechanism through the estrogenic and progestin action exerted by EE and NGM. The contraceptive effect of Effimia® is based on the interaction of various factors, the most important of which consist of ovulation inhibition and endometrial modifications.

SUMMARY:
As there are no recent studies conducted in Italy on the profile of this COC, the purpose of this study is to evaluate its efficacy and tolerability in a given subset of women residing in Italy that are in need of contraception. Evaluate the cycle control: breakthrough bleeding (bleeding and/or spotting between cyclically regular onset of menses) of monophasic oral contraceptive pill Effimia® (NGM250 + EE35) in a population of women residing in Italy.

ELIGIBILITY:
Inclusion Criteria:

* All the following criteria must be met.

  * Healthy women aged between 18 and 35 years (inclusive) in need of contraception.
  * Subjects residing in Italy and having a good knowledge of the Italian language, such as to correctly understand the Informed Consent Form, the instructions for use, and to ensure potential adhesion to the study.
  * Subjects providing written Informed Consent Form.
  * Subjects willing to comply with the study protocol.

Exclusion Criteria:

* Subjects who meet even one of the following criteria will be excluded from the study.

  * Subjects presenting any contraindications to the use of Combined Oral Contraceptives (COC) according to the current Summary of Product Characteristics (SmPC) of Effimia®, i.e. subjects presenting (or have ever presented) myocardial infarction, transient ischemic attack (TIA), stroke, angina pectoris, deep vein thrombosis (DVT), pulmonary embolism (PE) (or presence of blood clot in other organs than legs and lungs), any blood clotting disorder (such as protein C deficiency, protein S deficiency, antithrombin-III deficiency), or subjects that need to undergo surgery or that have to lie down for a long period of time (including the risk of previous deep vein thrombosis (DVT), arterial thromboembolism (ATE), hypertension in course of treatment and diabetes). If any of the listed conditions should appear during the use of the tested COC, the product must be stopped immediately, and the subject withdrawn from the study.
  * Subjects presenting severe diabetes with blood vessel damages, heart valve disease with complications, severe hypertension, severe hypercholesterolemia, or hypertriglyceridemia, hyperhomocysteinaemia, migraine with aura, hepatitis C (and taking medications for this condition), endometrial hyperplasia, unexplained vaginal bleeding, that are breastfeeding or pregnant or that are suspecting a pregnancy.
  * Subjects presenting (or have ever presented) any liver disease not yet recovered (liver function not yet normalized), any benign or malignant tumour of the liver, any breast or genital organs cancer (even suspected), jaundice during pregnancy or while using hormonal contraceptives.
  * Subjects presenting galactose intolerance, total lactase deficiency or glucosegalactose malabsorption syndrome.
  * Subjects presenting hypersensitivity to the active substances or to any excipients of the tested COC (e.g., norgestimate, ethinylstradiol or lactose).
  * Subjects using the following not allowed treatments during the whole study period (according to the SmPC of the Investigational Medicinal Product - IMP): treatments for tuberculosis (e.g. rifampicin), for epilepsy (e.g. primidone, phenytoin, barbiturates, carbamazepine, oxcarbazepine), for HIV and hepatitis C virus infection (protease inhibitor drugs and non-nucleoside reverse transcriptase inhibitors such as ritonavir, nevirapine, efavirenz and also ombitasvir, paritaprevir, ritonavir and dasabuvir), for fungal infections (e.g. griseofulvin), for arthritis, for osteoarthritis (etoricoxib ), for pulmonary arterial hypertension (bosentan) and St. John's wort used as an antidepressant. Medicines containing cyclosporine, the antiepileptic lamotrigine, tranexamic acid, theophylline (used to treat respiratory problems) and tizanidine (used to treat muscle pain and / or cramps) should not be taken as well.
  * Subjects who have used hormonal contraceptives in the previous month.
  * Subjects presenting a Body Mass Index - BMI ≥ 30 kg/m2 (class I obesity).
  * Subjects smoking > 15 cigarettes per day.
  * Subjects using COC off-label (e.g., for polycystic ovarian syndrome - PCOS, endometriosis, or recurrent menometrorrhagia).
  * Subjects currently taking part or who took part in clinical studies with experimental products in the previous month.
  * Subjects showing incapacity / inability to comply with the study protocol (unreliability in the intake of the product or in the completion of the diary) according to the Investigator's opinion.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy women aged between 18 and 35 years (inclusive) in need of contraception
Enrollment: 228 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Cycle control evaluation parameter | 180 days
  breakthrough bleeding (bleeding and/or spotting between cyclically regular onset of menses) by calculating the intermenstrual spotting occurrence rate at sixth cycle only (value to be intended as not cumulative with values from the other 5 cycles taking place during the whole study period). A comparison within group will be performed at V3 with respect to Baseline (V1)

SECONDARY OUTCOMES:
Cycle control evaluation parameters | 180 days
  frequency, duration, regularity, flow volume (subject determined), unscheduled bleeding. A comparison within group will be performed at V2 and V3 with respect to Baseline (V1).
Global Acne Grading System (GAGS). | 180 days
  A comparison within group will be performed at V2 and V3 with respect to Baseline (V1).
Profile of Mood State (POMS). | 180 days
  A comparison within group will be performed at V2 and V3 with respect to Baseline (V1).
Female Sexual Function Index (FSFI). | 180 days
  A comparison within group will be performed at V2 and V3 with respect to Baseline (V1).
Dysmenorrhea - VAS scale. | 180 days
  A comparison within group will be performed at V2 and V3 with respect to Baseline (V1)
Compliance | 180 days
  Adherence to treatment
Contraception failure rate during the 6-month treatment | 180 days
  the contraception failure rate is defined as the proportion of women who will become pregnant during the study period. The reasons for any contraception failure occurrence will be identified and listed (e.g., discontinuation or poor compliance).
Metabolic and hormonal parameters | 180 days
  blood lipid and glucose parameters (total cholesterol, High Density Lipoprotein - Cholesterol HDL-C, Low Density Lipoprotein - Cholesterol LDL-C, triglycerides, total testosterone, dehydroepiandrosterone - DHEAS, androstenedione, glucose, insulin, Sex Hormone Binding Globulin - SHBG) and hyperandrogenism (Free Androgenicity Index - FAI) - only in a subgroup of 28 subjects recruited only in the centre of Genova. They will be evaluated in comparison with Baseline (V1).

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Cagnacci, MD, Principal Investigator — IRCCS Ospedale Policlinico San Martino, Clinica Ostetrica e Ginecologica
Locations (1):
- IRCCS Ospedale Policlinico, San Martino, Genova, Italy

REFERENCES:
- [Background] Mosher WD, Martinez GM, Chandra A, Abma JC, Willson SJ. Use of contraception and use of family planning services in the United States: 1982-2002. Adv Data. 2004 Dec 10;(350):1-36. PMID 15633582
- [Background] Trussell J. Contraceptive failure in the United States. Contraception. 2011 May;83(5):397-404. doi: 10.1016/j.contraception.2011.01.021. Epub 2011 Mar 12. PMID 21477680
- [Background] Brynhildsen J. Combined hormonal contraceptives: prescribing patterns, compliance, and benefits versus risks. Ther Adv Drug Saf. 2014 Oct;5(5):201-13. doi: 10.1177/2042098614548857. PMID 25360241
- [Background] Sitruk-Ware R, Nath A. Characteristics and metabolic effects of estrogen and progestins contained in oral contraceptive pills. Best Pract Res Clin Endocrinol Metab. 2013 Feb;27(1):13-24. doi: 10.1016/j.beem.2012.09.004. Epub 2012 Oct 10. PMID 23384742
- [Background] European Medicines Agency Benefits of combined hormonal contraceptives (CHCs) continue to outweigh risks - CHMP endorses PRAC recommendation EMA/709120/2013 Available at: http://www.ema.europa.eu/ema/index.jsp?curl=pages/news_and_events/news/2013/11/news_d etail_001969.jsp&mid=WC0b01ac058004d5c1
- [Background] Phillips A, Hahn DW, McGuire JL. Preclinical evaluation of norgestimate, a progestin with minimal androgenic activity. Am J Obstet Gynecol. 1992 Oct;167(4 Pt 2):1191-6. doi: 10.1016/s0002-9378(12)90410-x. PMID 1415445
- [Background] Bottiger LE, Boman G, Eklund G, Westerholm B. Oral contraceptives and thromboembolic disease: effects of lowering oestrogen content. Lancet. 1980 May 24;1(8178):1097-101. doi: 10.1016/s0140-6736(80)91550-0. PMID 6103437
- [Background] Goldzieher JW. Selected aspects of the pharmacokinetics and metabolism of ethinyl estrogens and their clinical implications. Am J Obstet Gynecol. 1990 Jul;163(1 Pt 2):318-22. doi: 10.1016/0002-9378(90)90575-r. PMID 2196804
- [Background] Gallo MF, Nanda K, Grimes DA, Lopez LM, Schulz KF. 20 microg versus >20 microg estrogen combined oral contraceptives for contraception. Cochrane Database Syst Rev. 2013 Aug 1;2013(8):CD003989. doi: 10.1002/14651858.CD003989.pub5. PMID 23904209
- [Background] Van Vliet HA, Raps M, Lopez LM, Helmerhorst FM. Quadriphasic versus monophasic oral contraceptives for contraception. Cochrane Database Syst Rev. 2011 Nov 9;(11):CD009038. doi: 10.1002/14651858.CD009038.pub2. PMID 22071862
- [Background] Runnebaum B, Grunwald K, Rabe T. The efficacy and tolerability of norgestimate/ethinyl estradiol (250 micrograms of norgestimate/35 micrograms of ethinyl estradiol): results of an open, multicenter study of 59,701 women. Am J Obstet Gynecol. 1992 Jun;166(6 Pt 2):1963-8. doi: 10.1016/0002-9378(92)91396-r. PMID 1605286
- [Background] National Research Council (US) Committee on Population. Contraception and Reproduction: Health Consequences for Women and Children in the Developing World. Washington (DC): National Academies Press (US); 1989. Available from http://www.ncbi.nlm.nih.gov/books/NBK235072/ PMID 25144060
- [Background] Dayal M, Barnhart KT. Noncontraceptive benefits and therapeutic uses of the oral contraceptive pill. Semin Reprod Med. 2001 Dec;19(4):295-303. doi: 10.1055/s-2001-18637. PMID 11727171
- [Background] PASS 2021 Power Analysis and Sample Size Software (2021). NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass
- [Background] Doshi A, Zaheer A, Stiller MJ. A comparison of current acne grading systems and proposal of a novel system. Int J Dermatol. 1997 Jun;36(6):416-8. doi: 10.1046/j.1365-4362.1997.00099.x. No abstract available. PMID 9248884
- [Background] Alsulaimani H, Kokandi A, Khawandanh S, Hamad R. Severity of Acne Vulgaris: Comparison of Two Assessment Methods. Clin Cosmet Investig Dermatol. 2020 Sep 28;13:711-716. doi: 10.2147/CCID.S266320. eCollection 2020. PMID 33061511
- [Background] McNair, D. M., Lorr, M., & Droppleman, L. F. (1971). Manual for the Profile of Mood States. San Diego, CA: Educational and Industrial Testing Services.
- [Background] McNair, D. M., Lorr, M., & Droppleman, L. (1971/1981). Manual for the Profile of Mood States. San Diego, CA: Educational and Industrial Testing Service.
- [Background] McNair DM et al. Manual for the profile of Mood States. Toronto, ON, Multi-Health Systems Inc.1992.
- [Background] Evans SM, Haney M, Levin FR, Foltin RW, Fischman MW. Mood and performance changes in women with premenstrual dysphoric disorder: acute effects of alprazolam. Neuropsychopharmacology. 1998 Dec;19(6):499-516. doi: 10.1016/S0893-133X(98)00064-5. PMID 9803426
- [Background] Rapkin Andrea, L. H. Chang & A. E. Reading (1987) Premenstrual syndrome: a double blind placebo controlled study of treatment with progesterone vaginal suppositories, Journal of Obstetrics and Gynaecology, 7:3, 217-220, DOI: 10.3109/01443618709068522
- [Background] Wyatt K, Dimmock P, Jones P, Obhrai M, O'Brien S. Efficacy of progesterone and progestogens in management of premenstrual syndrome: systematic review. BMJ. 2001 Oct 6;323(7316):776-80. doi: 10.1136/bmj.323.7316.776. PMID 11588078
- [Background] Mannarini, S., Polimeni, S., Shams, M., & Giacobbo, M. (2012). Assessing negative and positive mood states: The identification of a short form of the POMS scale in Italian oncology outpatients. TPM - Testing, Psychometrics, Methodology in Applied Psychology, 19(2), 135- 145. https://doi.org/10.4473/TPM19.2.5
- [Background] Farnè, M., Sebellico, A., Gnugnoli, D., & Corallo, A. (1991). POMS: Profile Of Mood States. Adattamento italiano [POMS: Profile Of Mood States. Italian Adaptation]. Firenze, Italy: Organizzazioni Speciali.
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Wiegel M, Meston C, Rosen R. The female sexual function index (FSFI): cross-validation and development of clinical cutoff scores. J Sex Marital Ther. 2005 Jan-Feb;31(1):1-20. doi: 10.1080/00926230590475206. PMID 15841702
- [Background] Filocamo MT, Serati M, Li Marzi V, Costantini E, Milanesi M, Pietropaolo A, Polledro P, Gentile B, Maruccia S, Fornia S, Lauri I, Alei R, Arcangeli P, Sighinolfi MC, Manassero F, Andretta E, Palazzetti A, Bertelli E, Del Popolo G, Villari D. The Female Sexual Function Index (FSFI): linguistic validation of the Italian version. J Sex Med. 2014 Feb;11(2):447-53. doi: 10.1111/jsm.12389. Epub 2013 Nov 13. PMID 24224761
- [Background] Rosner W, Auchus RJ, Azziz R, Sluss PM, Raff H. Position statement: Utility, limitations, and pitfalls in measuring testosterone: an Endocrine Society position statement. J Clin Endocrinol Metab. 2007 Feb;92(2):405-13. doi: 10.1210/jc.2006-1864. Epub 2006 Nov 7. PMID 17090633
- [Background] Bhatt A. Protocol deviation and violation. Perspect Clin Res. 2012 Jul;3(3):117. doi: 10.4103/2229-3485.100663. No abstract available. PMID 23125964
- [Background] Ghooi RB, Bhosale N, Wadhwani R, Divate P, Divate U. Assessment and classification of protocol deviations. Perspect Clin Res. 2016 Jul-Sep;7(3):132-6. doi: 10.4103/2229-3485.184817. PMID 27453830
- [Background] Fraser IS, Critchley HO, Munro MG, Broder M; Writing Group for this Menstrual Agreement Process. A process designed to lead to international agreement on terminologies and definitions used to describe abnormalities of menstrual bleeding. Fertil Steril. 2007 Mar;87(3):466-76. doi: 10.1016/j.fertnstert.2007.01.023. PMID 17362717
- [Background] Fraser IS, Critchley HO, Munro MG, Broder M. Can we achieve international agreement on terminologies and definitions used to describe abnormalities of menstrual bleeding? Hum Reprod. 2007 Mar;22(3):635-43. doi: 10.1093/humrep/del478. Epub 2007 Jan 4. PMID 17204526
- [Background] Fraser IS, Critchley HO, Broder M, Munro MG. The FIGO recommendations on terminologies and definitions for normal and abnormal uterine bleeding. Semin Reprod Med. 2011 Sep;29(5):383-90. doi: 10.1055/s-0031-1287662. Epub 2011 Nov 7. PMID 22065325
- [Derived] Cagnacci A, Grandi G, Capobianco G, Fulghesu AM, Morgante G, Biondelli V, Piccolo E, Casolati E, Mangrella M. Effects of a Monophasic Hormonal Contraceptive With Norgestimate+Ethinyl Estradiol on Menstrual Bleeding: Protocol and Design of a Multicenter, Prospective, Open-Label, Noncomparative Study in Italy. JMIR Res Protoc. 2025 Mar 31;14:e63683. doi: 10.2196/63683. PMID 40164172